CLINICAL TRIAL: NCT06939543
Title: The Test of Those Managing Pain With Their Own Pain" - A Questionnaire-Based Study on Pain Perception and Patient Empathy Among Physicians Actively Managing Pain
Brief Title: The Test of Those Managing Pain With Their Own Pain
Status: Not yet recruiting | Type: Observational
Sponsor: Haseki Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Ali Hüseyin Demir, MD, Haseki Training and Research Hospital
Other Study IDs: HASEKİ ANKET İLKE HOCA
Record Dates: First submitted 2025-04-10; First posted 2025-04-23 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Empathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: empathy — physicians' awareness of their health status, empathy towards patients

SUMMARY:
The study aims primarily to investigate physicians' awareness of their health status, empathy towards patients, and management processes through a questionnaire targeting physicians who diagnose and manage patients' pain.

ELIGIBILITY:
Inclusion Criteria:

* Specialist physicians actively working in pain treatment and management (e.g., Algology, Physical Medicine and Rehabilitation, Anesthesiology, Neurology, Rheumatology, etc.) or physicians currently undergoing specialty training in these areas.
* Physicians who volunteer to participate in the study and sign the informed consent form.
* Physicians who have actively followed up patients and applied pain management techniques within the last year.

Exclusion Criteria:

* Physicians who are not actively involved in pain management or who specialize in different medical fields.
* Physicians who do not wish to complete the questionnaire or do not provide voluntary consent.
* Physicians who complete the questionnaire incompletely or invalidly during the study.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Physicians working in anesthesiology, algology, intensive care, neurology, and physical therapy.
Sampling Method: Non-Probability Sample
Enrollment: 175 (Estimated)
Dates: Start 2025-04-11 (Estimated); Primary Completion 2025-04-20 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
pain questionnaire | 1 week
  questionnaire ( no pain:1 and worst pain:5 )

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ruscheweyh R, Marziniak M, Stumpenhorst F, Reinholz J, Knecht S. Pain sensitivity can be assessed by self-rating: Development and validation of the Pain Sensitivity Questionnaire. Pain. 2009 Nov;146(1-2):65-74. doi: 10.1016/j.pain.2009.06.020. Epub 2009 Aug 7. PMID 19665301
- [Result] Licciardone JC, Tran Y, Ngo K, Toledo D, Peddireddy N, Aryal S. Physician Empathy and Chronic Pain Outcomes. JAMA Netw Open. 2024 Apr 1;7(4):e246026. doi: 10.1001/jamanetworkopen.2024.6026. PMID 38602675